CLINICAL TRIAL: NCT01270308
Title: Open Label, Randomized, Two-treatment, Three-period, Three-sequence, Partial Replicate Oral Bioequivalence Study of Lansoprazole 30 mg DR Capsules of Dr.Reddy's Laboratories Limited, India Comparing With That of PREVACID® (Containing Lansoprazole) 30 mg DR Capsules of TAP Pharmaceuticals Inc. USA, in Healthy, Adult, Human Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Lansoprazole DR Capsules 30 mg in Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Manager - Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-699/08
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: Bioequivalence; two way crossover
MeSH Terms: interventions — Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lansoprazole DR Capsules 30 mg (Experimental): Lansoprazole DR Capsules 30 mg of Dr.Reddy's Laboratories Limited
  Interventions: Drug: Lansoprazole
- Prevacid 30 mg Capsules (Active Comparator): Prevacid 30 mg Capsules of TAP Pharmaceuticals Inc. USA
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole — Lansoprazole DR Capsules 30 mg
  Other Names: Prevacid

SUMMARY:
The objective of this study was to compare the relative bioavailability of Lansoprazole DR Capsules 30 mg with Prevacid® Capsules 30 mg under fasting conditions in healthy adult human subjects.

DETAILED DESCRIPTION:
open label, randomized, two-treatment, three-period, three-sequence, partial replicate oral bioequivalence study of Lansoprazole 30 mg DR Capsules of Dr.Reddy's Laboratories Limited, India comparing with that of PREVACID® (containing Lansoprazole) 30 mg DR Capsules of TAP Pharmaceuticals Inc. USA, in healthy, adult, human subjects under fasting conditions. 48 healthy, adult, human subjects were enrolled in the study and 42 subjects were completed the study.

ELIGIBILITY:
Inclusion Criteria:

i. Provided written informed consent.

ii. Subject who were healthy, adult, human beings within 18 and 45 years of age (both inclusive) weighing at least 50 kg.

iii. Subject having a body mass index between 18.0 and 29.9 (both inclusive), calculated as weight in Kg/height in m2.

iv. Subject having a normal health as determined by medical history, physical examination and laboratory investigation performed within 28 days prior to the commencement of the study. (Laboratory values must be within normal limits or considered by the physician /investigator to be of no clinical significance).

v. Female Subjects of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence.

* postmenopausal for at least 1 year.
* surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject)

Exclusion Criteria:

i. Subject who were incapable of understanding the informed consent.

ii. Systolic blood pressure less than 90 mm of Hg or more than 140 mm of Hg.

iii. Diastolic blood pressure less than 60 mm of Hg or more than 90 mm of Hg.

iv. Oral temperature is below 95.0°F or above 98.6°F.

v. Pulse rate below 50/min or above 100/min.

vi. History of hypersensitivity or idiosyncratic reaction to investigational drug product or any other related drugs.

vii. Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function.

viii. Consumption of grapefruit for the past ten days prior to the check-in, in each period.

ix. Regular smoker who has a habit of smoking more than nine cigarettes per day and has difficulty in abstaining from smoking during sample collection period.

x. Habit of alcoholism and difficulty in abstaining from alcohol during the sample collection period.

xi. Difficulty in abstaining from xanthene containing food or beverages (like tea, coffee, chocolates and cola drinks) during the sample collection period.

xii. Intake of over the counter (OTC) or prescribed medications and enzyme modifying medication or systemic medication for the last 30 days before dosing.

xiii. Clinically significant abnormalities and / or with significant diseases.

xiv. Confirmed positive in alcohol screening.

xv. Confirmed positive in selected drug of abuse.

xvi. Subjects who had participated in any other clinical investigation using experimental drug/donated blood in past 90 days before the date of start of study

xvii. Confirmed positive in urine pregnancy test.

xviii. Female detected to be pregnant, breast feeding or who is likely to become pregnant during the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr.M.Venkat Jayanth, MBBS, Principal Investigator — Bioserve Clinical Research (P) Ltd
Locations (1):
- Bioserve Clinical Research (P) Ltd, Bālānagar, Hyderabad, India